CLINICAL TRIAL: NCT06294678
Title: A Multicenter Randomized Controlled Study of the Effect of Stem Cell Infusion Time on the Development of aGVHD in Patients With Hematological Malignancies After Allogeneic Peripheral Blood Hematopoietic Stem Cell Transplantation
Brief Title: Effect of Stem Cell Infusion Time on aGVHD in Patients With Hematological Malignancies
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: infusion time & aGVHD-001
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Graft-versus-host Disease
Keywords: Time of stem cell infusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the early infused group (Active Comparator): infused stem cell within 11:30 am and 12:30 am
  Interventions: Procedure: Time of stem cell infusion
- the late infused group (Sham Comparator): infused stem cell within 5:30 pm and 6:30 pm
  Interventions: Procedure: Time of stem cell infusion

INTERVENTIONS:
Procedure: Time of stem cell infusion — Randomization of patients according to the time of stem cell infusion

SUMMARY:
To observe the effect of stem cell infusion on the development of acute graft-versus-host disease (aGVHD) in patients with malignant hematologic diseases after allogeneic peripheral blood hematopoietic stem cell transplantation (allo-PBSCT)

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGVHD) is a major complication and non-recurrent cause of death after allogeneic hematopoietic stem cell transplantation (allo-HSCT). The human biological clock uses recurring environmental cues such as light and food intake to establish 24-hour rhythmic changes in sleep, hormone secretion, metabolism, body temperature, and immune function. Current clinical aGVHD prevention strategies focus on suppression of donor lymphocyte function by drugs or immunomodulatory cells, ignoring the impact of the recipient's own functional changes on the graft. The applicant's previous retrospective cohort study found that the time of stem cell infusion severely affected the incidence of aGVHD and its severity after allogeneic peripheral blood hematopoietic stem cell transplantation (allo-PBSCT). Due to the lack of prospective clinical trial results on the effect of stem cell infusion time on the occurrence of aGVHD after allo-HSCT in the international arena, as well as the possible influence of multiple confounding factors in the aforementioned single-center retrospective study, the present study intends to randomize patients according to the time of stem cell infusion, and to observe its effect on the incidence of aGVHD, other transplant-related complications, and long-term survival after allo-PBSCT of patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of malignant hematologic disease before transplantation, age 12-60 years old, gender is not limited, race is not limited;
* Patients who are proposed to receive allo-PBSCT for the first time;
* Eastern Cooperative Oncology Group (ECOG) score 0-2;
* No serious organ failure and active infection;
* Voluntary open randomized controlled study to observe whether the time of stem cell infusion affects the occurrence of aGVHD after transplantation;
* Each subject must sign an informed consent form (ICF) indicating that he/she understands the purpose and procedures of the study and is willing to participate in the study; in view of the patient's condition, if the patient's own signature is not conducive to the treatment of his/her condition, the ICF will be signed by the legal representative.

Exclusion Criteria:

* Those with severe organ dysfunction or disease, such as severe disease and dysfunction of the heart, liver, kidneys and pancreas;
* Pregnant patients;
* Patients and/or authorized family members who refuse to undergo an open randomized controlled study to observe whether the time of stem cell infusion affects the occurrence of aGVHD after transplantation;
* Any life-threatening disease, physical condition, or organ system dysfunction that, in the opinion of the investigator, may compromise patient safety and put the results of the study at unnecessary risk; drug-dependent individuals; patients with uncontrolled psychiatric disorders; and individuals with cognitive dysfunction;
* Participants in other clinical studies that may affect aGVHD within 3 months;
* Those whom the investigator considers unsuitable for enrollment (e.g., those who anticipate that patients will not be able to adhere to the examination and treatment due to financial and other issues).

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade II to IV aGVHD | 100 days
  The primary endpoint of the study will be the development of grade II to IV aGVHD in the first 100 days post-transplant. Acute GVHD was graded according to the Mount Sinai Acute GVHD International Consortium criteria.

SECONDARY OUTCOMES:
The incidence of grade III to IV aGVHD | 100 days
  The cumulative incidence of grade III to IV aGVHD in the first 100 days post-transplant. aGVHD was graded according to the Mount Sinai Acute GVHD International Consortium criteria.
The cumulative incidence of neutrophil engraftment at 28 days after transplantation | 28 days
  neutrophil engraftment time was defined as the first of three consecutive days during which the neutrophil count was at least 0.5×10^9/L.
The cumulative incidence of platelet recovery at 100 days after transplantation | 100 days
  Platelet recovery is defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥ 100 × 10^9/L.
The cumulative incidence of transplant-related mortality at 180 days after transplantation | 180 days
  The cumulative incidence of transplant-related mortality at 180 days after transplantation
The cumulative incidence of transplant-related mortality at 360 days after transplantation | 360 days
  The cumulative incidence of transplant-related mortality at 360 days after transplantation
The cumulative incidence of chronic GVHD at 360 days after transplantation | 360 days
  The severity of chronic GVHD was graded according to the 2014 NIH criteria.
The probability of GVHD-free, relapse-free survival(GRFS) | 360 days
  The composite endpoint of GRFS was defined as the first events occurring after transplantation among Grade III to IV aGVHD, moderate to severe cGVHD, relapse, or death for any reason.
The probability of disease-free survival(DFS) | 360 days
  The DFS was defined as the interval between transplantation and disease recurrence, death or the last follow-up date, whichever occurred first.
The probability of overall survival(OS) | 360 days
  The OS was determined to be the time from the first day of transplantation until death from any cause or the last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, ph.D, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (6):
- China (6):
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Rui Jin Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No